- 1 RELIABILITY AND VALIDITY OF THE INTERNATIONAL STANDARDS FOR
- 2 NEUROLOGICAL CLASSIFICATION OF SPINAL CORD INJURY IN PATIENTS WITH
- 3 NON-TRAUMATIC SPINAL CORD LESIONS

4

- 5 PROJECT
- 6 PATIENTS AND METHODS
- 7 All patients with non-traumatic SCI consecutively admitted to three Italian SCI centers (IRCCS
- 8 Fondazione Santa Lucia, Montecatone Rehabilitation Hospital and Istituti Clinici Scientifici
- 9 Maugeri IRCCS of Pavia) between January 1<sup>st</sup> 2017 and June 30<sup>th</sup> 2020 have been prospectively
- 10 enrolled in the study.
- 11 The study has been registered at Clinicatrials.gov.
- 12 The study was approved by the ethic committee of IRCCS Fondazione Santa Lucia and all the
- patients signed an informed consent to the study.
- Inclusion criteria were: having a non-traumatic SCI in the acute / subacute phase with any level and
- severity (ASIA Impairment Scale) of injury and having a cognitive status that allows collaboration
- in the exam.
- Exclusion criteria were the presence of dementia or cognitive decline; having a pathology of the
- peripheral nervous system that may affect the evaluation of ISNCSCI; having a multiple sclerosis.
- 19 The following data were prospectively recorded:
- Recording of demographic and clinical history data. Concerning the onset of lesion, for the
- 21 ischemic and inflammatory groups reference was made to the appearance of the first symptoms,

- 22 while for the neoplastic and spondylogenetic myelopathies we referred to the date of surgical
- 23 intervention which is usually accompanied by a worsening of the clinical picture.
- Evaluation of neurological conditions according to the International Standards For Neurological
- Classification of Spinal Cord Injury (ISNCSCI) (Revision 2015) (23) with registration of right and
- left motor and sensory level and of the Neurological Level of Injury (NLI), of the total motor score
- 27 (MS), of upper extremities (UEMS) and lower extremities (LEMS) motor scores, light touch and
- 28 pin prick sensory scores, and ASIA Impairment Scale (AIS). This assessment was carried out by
- 29 two different experienced examiners (Table 1) in each center, 48-72 hours apart. One of the two
- 30 examiners also assessed the functional status of the patients through the Spinal Cord Independence
- 31 Measure (SCIM) version 2 or 3 (24).
- The patients were evaluated at admission with the possibility of repeating the evaluation also
- during rehabilitation stay and at discharge,.

- 34 Statistics
- 35 Descriptive statistics: mean and standard deviation (SD) for quantitative data; frequencies and
- 36 percentages for qualitative ones. Normality of data was assessed by Shapiro-Wilk test. The NLI and
- 37 the AIS grade have been transformed into numbers and treated as ordinal variables. For the NLI the
- level C1 corresponds to 1, and the level S4-5 to the number 29. For the AIS grade A correspond to 1
- and grade E to 5.
- 40 Validity and reliability represents the main measurement psychometric properties of instruments.
- The validity of instrument means that it measures what it is intended to measure. (25) while
- reliability refers to its stability over time (26).
- Different aspects of reliability were assessed with appropriate tests: correlation (Spearman), test-
- retest reliability (Krippendorf's Alpha) and internal consistency (Cronbach's Alpha) (27, 28). For
- 45 motor and sensory scores, we also compared the data of the two examiners by means of Wilcoxon
- 46 matched pair test to evaluate if there was any significant difference.
- As to the levels of injury (Neurological Level of Injury, left and right sensory and motor level of
- 48 injury) and AIS grade the agreement between the two examiners regarding was assessed through the
- 49 Krippendorff's Alpha. Furthermore, for the assessment of the levels, we compared the levels
- established by the two examiners, by counting the difference (1 level, 2 or move levels) in cases
- 51 where assessments differed.
- We evaluate psychometric properties of AIS scale on all sample and in each pathology subgroups.
- As currently there is no gold standard for the neurological evaluation of persons with SCI other than
- 54 the ISNCSCI, we have evaluated the convergent construct validity of the Standards through a
- 55 Spearman correlation between the total motor scores, the upper and lower extremities motor scores
- and the total SCIM score as well as the subscores "Self-care" and "Mobility". This correlation was
- 57 performed by means of Spearman test.

- According to Landis and Koch (29), we interpreted ICC values and the level of agreement by
- 59 Kappa-values as follows:
- 60 0–0.1-virtually none
- 61 0.1–0.4-slight
- 62 0.41–0.6-fair
- 63 0.61–0.8-moderate
- 64 0.81–1-substantial
- All analyses were performed with SPSS 22.
- 66 Significance was set at p<0.05
- Data have been reported according to the Guidelines For Reporting Reliability And Agreement
- 68 Studies (GRRAS) (supplemental material, Table 15).